CLINICAL TRIAL: NCT00002111
Title: A Dose-Escalating Study of Ro 31-8959 ( HIV Protease Inhibitor ) in Patients With HIV Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 212A; EV 14757
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-05

CONDITIONS: HIV Infections
Keywords: AIDS-Related Complex; Saquinavir; HIV Protease Inhibitors
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Saquinavir

INTERVENTIONS:
Drug: Saquinavir

SUMMARY:
To investigate the toxicity, antiviral activity, and pharmacokinetics in HIV-infected patients receiving 16 weeks of oral saquinavir mesylate ( Ro 31-8959 ) at one of two doses.

DETAILED DESCRIPTION:
Cohorts of 16 patients receive 1 of 2 doses of Ro 31-8959 for 20 weeks. Administration of the higher dose will proceed only after 2-week safety data for the first eight patients on the lower dose has been reviewed.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV infection.
* CD4 count 200 - 500 cells/mm3.
* No evidence of viral resistance.
* HIV RNA quantifiable by PCR.
* Negativity for HBsAg, HBeAg, and anti-HBc.

NOTE:

* Fifty percent of patients must have measurable p24 antigen levels (> 31 pg/ml).

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active opportunistic infection requiring immediate treatment, such as tuberculosis, cytomegalovirus, cerebral toxoplasmosis, and Pneumocystis carinii pneumonia.
* Unable to maintain adequate oral intake.
* Clinically significant vomiting and/or diarrhea.
* Malignancy, visceral Kaposi's sarcoma, or lymphoma that will require systemic chemotherapy within the next 12 months.
* Unable to comply with protocol requirements, in the judgment of the investigator.
* Any grade 3 or worse laboratory or clinical abnormality.

Concurrent Medication:

Excluded:

* Antineoplastic agents.
* Concomitant or maintenance treatment with excluded experimental drugs and drugs with known nephrotoxic or hepatotoxic potential.

Concurrent Treatment:

Excluded:

* Radiation therapy other than local skin radiation therapy.

Patients with the following prior conditions are excluded:

* Unexplained temperature >= 38.5 C (101.5 F) persisting for 14 days or more within a 30-day period.
* Unexplained, chronic diarrhea persisting for 14 days or more within a 30-day period.

Prior Medication:

Excluded:

* Prior treatment with an HIV proteinase inhibitor.
* AZT within 30 days prior to study entry OR lasting more than 1 year.
* Other antiretroviral therapy (besides AZT) within 30 days prior to study entry OR lasting more than 14 days.
* Acute therapy for an opportunistic infection within 14 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Univ School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Schapiro JM, Winters MA, Stewart F, Efron B, Norris J, Kozal MJ, Merigan TC. The effect of high-dose saquinavir on viral load and CD4+ T-cell counts in HIV-infected patients. Ann Intern Med. 1996 Jun 15;124(12):1039-50. doi: 10.7326/0003-4819-124-12-199606150-00003. PMID 8633817